CLINICAL TRIAL: NCT03976882
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Hetrombopag in Subjects With Chemotherapy-induced Thrombocytopenia Receiving Chemotherapy for the Treatment of Solid Tumors.
Brief Title: Hetrombopag for the Treatment of Chemotherapy-Induced Thrombocytopenia in Subjects With Malignancy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-TPO-CIT-III
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Chemotherapy-Induced Thrombocytopenia
MeSH Terms: interventions — hetrombopag

STUDY DESIGN:
Intervention Model Description: Hetrombopag compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A：Hetrombopag (Experimental)
  Interventions: Drug: Hetrombopag
- Group B：Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hetrombopag — Hetrombopag
  Arms: Group A：Hetrombopag
Drug: Placebo — Placebo
  Arms: Group B：Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of Hetrombopag in subjects with chemotherapy-induced thrombocytopenia receiving chemotherapy for the treatment of solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, 18-75 years of age;
2. Participant with a confirmed diagnosis of solid tumor receiving a chemotherapy regimen;
3. Participant experienced thrombocytopenia and chemotherapy delay;
4. ECOG performance status 0-1;

Exclusion Criteria:

1. Screening and baseline platelet count< 30×109/L;
2. Participant has experienced thrombocytopenia due to any etiology other than chemotherapy within 6 months of screening;
3. Participant has any history of hematologic diseases other than chemotherapy-induced thrombocytopenia;
4. Participant has serious bleeding symptoms;
5. Participant has no hepatic metastases, ALT/AST>3ULN, TBIL>3ULN; with hepatic metastases, ALT/AST≥5ULN, TBIL≥5ULN;
6. Blood Cr≥1.5ULN or eGFR≤60 ml/min（Cockcroft-Gault）;
7. History of allergy to the study drug;
8. Participant with HIV;
9. Pregnant or lactating women;
10. Other conditions that may affect participant's safety or trial evaluations per investigator's discretion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
The proportion of treatment responders. | Randomization up to 90 days

SECONDARY OUTCOMES:
Duration from starting treatment to initiating chemotherapy and platelet count ≥100×109/L | Randomization up to 30 days
Proportion of subjects who can completion chemotherapy without rescue therapy and dose modification | Randomization up to 150 days
Proportion of subjects without serious bleeding event | Randomization up to 180 days
Number of subjects with any Adverse Event (AE) or Serious Adverse Event (SAE) graded by the investigator according to National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE), version 5.0 | Randomization up to 180 days

CONTACTS AND LOCATIONS:
Locations (1):
- Najing Bayi Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Qin S, Wang Y, Yao J, Liu Y, Yi T, Pan Y, Chen Z, Zhang X, Lu J, Yu J, Zhang Y, Cheng P, Mao Y, Zhang J, Fang M, Zhang Y, Lv J, Li R, Dou N, Tang Q, Ma J. Hetrombopag for the management of chemotherapy-induced thrombocytopenia in patients with advanced solid tumors: a multicenter, randomized, double-blind, placebo-controlled, phase II study. Ther Adv Med Oncol. 2024 Jun 14;16:17588359241260985. doi: 10.1177/17588359241260985. eCollection 2024. PMID 38882443